CLINICAL TRIAL: NCT07044323
Title: Efficacy and Mechanisms of Virtual Reality Treatment of Phantom Leg Pain.Home-Based Treatment
Acronym: PLP Home-Based
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Laurel Buxbaum, Principal Investigator, Albert Einstein Healthcare Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEHN2022-775; 5R01HD104158-03 (NIH)
Record Dates: First submitted 2025-06-23; First posted 2025-06-30 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Phantom Pain Following Amputation of Lower Limb; Amputation
Keywords: pain; phantom limb; lower limb amputation; treatment
MeSH Terms: conditions — Pain; Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based treatment (Experimental): Self-administered Active Virtual Reality treatment
  Interventions: Behavioral: Active Virtual Reality Treatment

INTERVENTIONS:
Behavioral: Active Virtual Reality Treatment — The self-administered active VR treatment will consist of 8 twice-weekly sessions, each approximately 1 hour in duration, during which subjects will participate in a variety of Virtual Reality active games that require leg movements while receiving high-quality visual feedback of the missing lower leg.

SUMMARY:
After amputation of an arm or leg, up to 90% of subjects experience a "phantom limb", a phenomenon characterized by persistent feelings of the missing limb. Many subjects with a phantom limb experience intense pain in the missing extremity that is often poorly responsive to medications or other interventions. The study will explore the feasibility and efficacy of a home-based, active VR treatment for phantom limb pain (PLP).

DETAILED DESCRIPTION:
Almost 2 million people in the US have had an amputation and up to 90% of people with limb amputation experience the persistent sensation of the missing extremity, a phenomenon known as a "phantom limb"Additionally, a significant proportion of individuals with a phantom limb - up to 85% in some studies - experience persistent and debilitating pain in the missing limb, a condition known as phantom limb pain (hereafter PLP). Although existing therapies provide pain relief in some cases, there is widespread agreement that current approaches fall short of bringing relief to most individuals with PLP

The investigators recently completed the in-person part of the study in which they compared the efficacy of Active VR treatment to Distractor VR treatment for PLP on measures of pain as well as psychological health and quality of life.

In the Active VR treatment, subjects played a variety of active games requiring leg movements while receiving high-quality visual feedback of the missing lower leg. Feedback about leg position was provided via the VR headset controller, and the program generated an image of the missing lower leg, visible as a first-person avatar. The "Distractor" treatment was the REAL i-Series® immersive VR experience: subjects navigated through a pleasant VR environment, without seeing any rendering of their body and making no movements with their legs. The results of the in-person study showed superior efficacy in reducing pain intensity of the Active Treatment as compared to the Distractor treatment.

The specific aim of the current study is to assess the feasibility and efficacy of a home-based, active VR treatment for PLP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 -100
* Capacity to provide Informed Consent
* Unilateral above or below knee amputation more than 3 months prior to enrollment
* Absence of cognitive impairment, operationally defined as a Montreal Cognitive Assessment score of 18 or greater1.
* Pain averaged over the preceding 1 month in the phantom limb rated as greater than 4 on a scale of 0-10.

Exclusion Criteria:

* History of significant medical or neurological disorder such as stroke or moderate to severe traumatic brain injury (operationally defined as loss of consciousness for more than 30 minutes)
* History of significant or poorly controlled psychiatric disorders
* Substantial depression or anxiety affecting their ability to perform tasks necessary for the study.
* Current abuse of alcohol or drugs, prescription or otherwise
* Nursing a child, pregnant, or intent to become pregnant during the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes in pain intensity | pre each intervention (8 sessions); immediately after each intervention (8 session); baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention.
  the change in phantom limb pain score pre and post each VR intervention, at baseline, after the VR intervention and in the follow-up sessions as assessed using an 11-point numerical rating pain scale (0 - minimum score/no pain; 10 maximum score/pain as bad as you can imagine) assessing the current PLP level.
Changes in pain quality of the McGill Short Form Questionnaire | baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention
  The change in the phantom limb pain quality between baseline, post-intervention, and follow-up sessions using McGill Short Form Questionnaire that measures the characteristics of pain (e.g., throbbing, etc.) using a 4-point rating pain scale (0 - minimum score - none: better outcome /4 maximum score - severe: worse outcome).

SECONDARY OUTCOMES:
Changes in average pain after the treatment | up to 4 weeks
  average pain intensity since the previous intervention on an 11-point numerical rating pain scale; (0 - minimum score/no pain; 10 maximum score/pain as bad as participants can imagine); higher scores indicate higher level of pain (worse outcome)

OTHER OUTCOMES:
Changes in daily activities after the treatment | baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention
  The Frenchay Activities Index (FAI): a scale measuring the physical function and daily activity that has excellent reliability in subjects with lower-limb amputation in predicting quality of life. 0 minimum score - 45 maximum score; higher scores indicate more daily activities (better outcome).
Changes in quality of life after the treatment | baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention
  The 12-Item Short Form Health Survey (SF-12): a brief measure of quality of life and functional capacity that has been validated in patients with amputation and PLP. 0 minimum score - 100 maximum score. Higher scores indicate lower physical and mental health (worse outcome).
Changes in pain interference after the treatment | baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention
  The Pain Interference Scale from the Brief Pain Inventory (BPI): this assesses the degree to which pain interferes with daily activities using a 0-10 numeric rating scale. 0 minimum score - 10 maximum score. Higher scores indicate higher pain interference (worse outcome).
Changes in depression and anxiety as effect of the treatment | baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention
  The Hospital Anxiety and Depression Scale (HADS): the HADS is a 14- item measure assessing both depressive and anxiety symptoms. In addition to providing separate scores for anxiety and depression, the HADS also provides a measure of global negative affect. 0 minimum score - 42 maximum score. Higher scores indicate more depression and anxiety (worse outcome)
Changes in the pain catastrophizing after the treatment | baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention
  The 13-item Pain Catastrophizing Scale: this scale investigates pain catastrophizing, which has been highly associated with pain severity and disability after amputation. 0 minimum score -52; Higher scores indicate higher tendency to catastrophizing (worse outcome)
Changes in insomnia after the treatment | baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention
  Insomnia Severity Index: this is a 7-point scale that measure insomnia, a symptom associated with PLP. 0 minimum score - 28 maximum score; higher scores indicate more insomnia (worse outcome)
Perception of VR system | baseline, pre-intervention
  Technology Acceptance Scale (Morris et al., 1997): this is a 7-point scale that measure level of acceptance of the VR system. 0 minimum score - 133 maximum score; higher scores indicate low level of acceptance (worse score)
Usability of each game | immediately after the last intervention (session 8 of the intervention);
  System Usability Scale (SUS): Scale measuring the usability of each game; minimum score 10 - maximum score 50. Higher scores indicate less usability (worse outcome).
Simulator Sickness Questionnaire | day 1, day 8
  Simulator Sickness Questionnaire, which test for the presence of symptoms of cybersickness (e.g., general discomfort) on a 4-point numerical rating scale (0 - minimum score/no symptom; 4 maximum score/severe symptom)
Presence in VR | day 1, day 8
  Brief Slater-Usoh-Steed Presence Questionnaire. 7 minimum score - 42 maximum score. Higher scores indicate more presence in the VR (better outcome)
Changes in Phantom Limb and Phantom Limb Pain after the treatment | baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention
  The Modified Limb Deficiency and Phantom Limb Questionnaire: this questionnaire assesses the usage of prosthesis (yes/no) and non-painful phantom limb experiences (presence/absence), including perceived position (e.g., presence/absence of telescoping) and ability to move the phantom (yes/no).
Treatment satisfaction | 1 week after the end of the intervention
  visual analogue scale that evaluates treatment satisfaction; 0 minimum score - 10 maximum score; Higher scores indicate more treatment satisfaction (better outcome)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Jefferson Moss Rehabilitation Research Institute, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Slater M, Steed A, McCarthy J, Maringelli F. The influence of body movement on subjective presence in virtual environments. Hum Factors. 1998 Sep;40(3):469-77. doi: 10.1518/001872098779591368. PMID 9849105
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Goller AI, Richards K, Novak S, Ward J. Mirror-touch synaesthesia in the phantom limbs of amputees. Cortex. 2013 Jan;49(1):243-51. doi: 10.1016/j.cortex.2011.05.002. Epub 2011 Jun 22. PMID 22981809
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Holbrook M, Skilbeck CE. An activities index for use with stroke patients. Age Ageing. 1983 May;12(2):166-70. doi: 10.1093/ageing/12.2.166. PMID 6869117
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870